CLINICAL TRIAL: NCT06268145
Title: An Open-Label, Randomized, Single Dose, Crossover Clinical Study to Assess the Relative Bioavailability of Current Tablet Formulation (F1) Compared to New Tablet Formulation (F2) of ECC5004 and Food Effects on F1 and F2 of ECC5004 in Healthy Participants
Brief Title: ECC5004 RBA FE Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eccogene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EC0006
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fixed Sequence 1 (Experimental): Participants will receive single dose of ECC5004 F1 at fasted state, followed by F2 at fasted state, F1 at fed state and F2 at fed state in four treatment periods.
  Interventions: Drug: ECC5004
- Fixed Sequence 2 (Experimental): Participants will receive a single dose of ECC5004 F2 at fasted state, followed by F1 at fasted state, F2 at fed state, and F1 at fed state with four treatment periods.
  Interventions: Drug: ECC5004

INTERVENTIONS:
Drug: ECC5004 — A single dose tablet of 50 mg of the current tablet formulation (F1) or new tablet formulation (F2) administered orally.

SUMMARY:
This study is a Phase 1, open-label, randomized, single dose, fixed sequence, crossover study designed to compare the relative bioavailability of 50 mg ECC5004 current tablet formulation (F1) and 50 mg ECC5004 new tablet formulation (F2) under fasted and fed conditions in healthy participants

DETAILED DESCRIPTION:
Eligible participants will be randomized to one of the two fixed treatment sequences with four treatment periods. In the first two treatment periods under fasted conditions, participants will fast for a minimum of 10 hours, then they will receive a single dose of 50 mg ECC5004 F1 or 50 mg ECC5004 F2. In the subsequent third and fourth treatment periods under fed conditions, participants will consume completely a high fat breakfast followed by administration of a single dose of 50 mg ECC5004 F1 or 50 mg ECC5004 F2

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants of non-childbearing potential
* Age of 18 to 65 years
* BMI of 18.0 to 32.0 kg/m2
* Female participants who are postmenopausal, confirmed by FSH test, or surgically sterile, confirmed by medical documentation, or agree to practice true abstinence
* Male participants agree to use contraception, or agree to practice true abstinence
* No clinically significant findings in physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, clinical laboratory evaluations, concomitant medications, or medical/psychiatric history
* Able to understand and sign and date informed consent

Exclusion Criteria:

* Females who are pregnant, planning to become pregnant, or breastfeeding during the study or within 3 months after the study.
* Concomitant participation in any investigational study of any nature
* Blood loss of non-physiological reasons ≥ 200 ml (i.e. trauma, blood collection, blood donation) within 2 months prior to the first dose of study drug, or plan to donate blood during this trial and within 1 month after the last dosing
* Serum calcitonin > 20 ng/L
* Clinically relevant acute or chronic medical conditions or diseases of the cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric, immune or dermatologic systems
* Individual or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia 2 (MEN2), or suspected MTC
* History of pancreatitis
* Significant allergic reaction to active ingredients or excipients of the study drug
* Any clinically significant abnormal findings in the participant's physical examination, laboratory tests, pregnancy test, urine drug screen, alcohol test, or medical history which in the opinion of the Investigator would prevent the participants from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
ECC5004 PK parameters: AUC0-tlast | Up to day 6
  Area under the Plasma Concentration-Time Curve from Time 0 to the Last Measurable Non-Zero Concentration
ECC5004 PK parameters: AUC0-inf | Up to day 6
  Area under the Plasma Concentration-Time Curve from Time 0 Extrapolated to Infinity
ECC5004 PK parameters: Cmax | Up to day 6
  Maximum observed plasma concentration
ECC5004 PK parameters: tmax | Up to day 6
  Time of the maximum observed plasma concentration

SECONDARY OUTCOMES:
Number of participants with adverse events, with abnormal laboratory test results, abnormal ECGs, abnormal vital signs, and abnormal physical examinations | Up to Day 6
  Safety Assessment evaluated through adverse events, laboratory evaluations, vital signs, ECGs, and physical examination.
ECC5004 PK parameters: AUC0-tau | Up to day 6
  Area under the Plasma Concentration-Time Curve during the Dosing Interval
ECC5004 PK parameters: AUC 0-24 | Up to day 6
  Area under the Plasma Concentration-Time Curve from Time 0 to 24 Hours Post-dose
ECC5004 PK parameters: tlag | Up to day 6
  Lag time (time delay between dosing and first observed plasma concentration)
ECC5004 PK parameters: t1/2 | Up to day 6
  Apparent terminal elimination half-life
ECC5004 PK parameters: CL/F | Up to day 6
  Apparent Clearance
ECC5004 PK parameters: AUC(extr) | Up to day 6
  Area under the curve from the first measured concentration value back extrapolated to the concentration value at time zero as a percentage of the area under the curve extrapolated to infinity using the predicted value of the last non-zero concentration

CONTACTS AND LOCATIONS:
Overall Officials: Eccogene, Study Director — Eccogene Clinical Trials
Locations (1):
- Eccogene Investigational Site, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No